CLINICAL TRIAL: NCT05910645
Title: Knowledge, Attitude and Practice Regarding Caries Risk Assessment for Children and Adults Among Dental Residents :A Cross Sectional Study
Brief Title: Knowledge, Attitude and Practice Regarding Caries Risk Assessment for Children and Adults Among Dental Residents
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Manar Ramadan Ahmed Orabi, Doctor at Egyptian Ministry of Health, Cairo University
Other Study IDs: Caries Risk Assessment
Record Dates: First submitted 2023-06-01; First posted 2023-06-20 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Dental Residents in pediatric department
- Dental Residents in conservative department

SUMMARY:
Evaluation of knowledge, practice and attitude regarding Caries Risk Assessment for children and adults among Dental Residents in Faculty of Dentistry, Cairo University.

DETAILED DESCRIPTION:
Dental caries is a dynamic and multifactorial process. Occurrence of dental caries is affected by several factors including quantity and composition of saliva, oral microflora and patient-related parameters including general health and lifestyle, such as the use of fluoride-containing toothpastes and diet.

Caries risk is defined as the probability of developing caries in the future. The incidence of the disease can be either primary (New caries lesions) or secondary (Progression of lesion or reactivation of caries lesions). Caries risk assessment (CRA) is important for the successful application of a minimum intervention dentistry philosophy in the management of dental caries. Patients, with active caries at the time of visit, need the CRA to identify the factors that are most likely to progress in the disease process. The CRA is one of the methods for managing the caries of patients.

Riley et al. showed that the anti-caries agents were widely used in dental clinics, while the CRA was performed by a few dental clinics. In a study of Gaskin et al., 63.5% of subjects agreed with the use of minimal intervention dentistry. In a study of Shah et al., 36% of dentists accepted the use of restorative materials and CRA-based methods, and 15.5% also strongly agreed with CRA for all patients. In a study by Rayapudi and Usha, 81% of participants agreed with CRA in patients. In a study by Riley et al. about the use of CRA by dentists in children, 73% of dentists reported having CRAs for people aged 6 to 18 years. In another study by Riley et al., 69% of dentists performed CRA for patients, and 57% of dentists who performed CRA had considered an individualized caries prevention programs for their patients. Hurlbutt et al. showed that caries management by the CRA is an example of patient care that has the best practice rather than traditional therapies.

Afshar et al. claimed that the CRA is a conservative approach that can prevent waste of time, energy and finances. Evaluating the management of the results of illness in certain periods of time leads to less dental tissues wasting. People's knowledge of CRA in patients leads to more conservative treatment. Due to limited studies in this field and the absence of data about using CRA in Egypt, Especially on dental residents, this study was conducted to evaluate the knowledge, attitude and practice regarding Caries Risk Assessment among pediatric and Conservative Dental Residents in Faculty of Oral and Dental Medicine, Cairo University.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric and conservative dental residents in Faculty of Dentistry, Cairo University.

Completing at least 3 months residency program in one of the departments

Exclusion Criteria:

* Participants who refuse to participate.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: P1: Pediatric Dentistry Residents. P2: Conservative Dentistry Residents.
Sampling Method: Probability Sample
Enrollment: 3 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Knowledge regarding Caries Risk Assessment among Dental Residents in Faculty of Dentistry, CU Attitude regarding CRA among Dental Residents in Faculty of Dentistry, CU Practice regarding CRA among Dental Residents in Faculty of Dentistry, CU | through study completion, an average of 1 year
  Questionnaire Questionnaire Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Frencken JE, Peters MC, Manton DJ, Leal SC, Gordan VV, Eden E. Minimal intervention dentistry for managing dental caries - a review: report of a FDI task group. Int Dent J. 2012 Oct;62(5):223-43. doi: 10.1111/idj.12007. PMID 23106836
- [Background] Marsh PD. Microbiology of dental plaque biofilms and their role in oral health and caries. Dent Clin North Am. 2010 Jul;54(3):441-54. doi: 10.1016/j.cden.2010.03.002. PMID 20630188
- [Background] Hallett KB. The application of caries risk assessment in minimum intervention dentistry. Aust Dent J. 2013 Jun;58 Suppl 1:26-34. doi: 10.1111/adj.12047. PMID 23721335
- [Background] Twetman S, Fontana M. Patient caries risk assessment. Monogr Oral Sci. 2009;21:91-101. doi: 10.1159/000224214. Epub 2009 Jun 3. PMID 19494677
- [Background] Riley JL 3rd, Gordan VV, Rindal DB, Fellows JL, Ajmo CT, Amundson C, Anderson GA, Gilbert GH; Dental PBRN Collaborative Group. Preferences for caries prevention agents in adult patients: findings from the dental practice-based research network. Community Dent Oral Epidemiol. 2010 Aug;38(4):360-70. doi: 10.1111/j.1600-0528.2010.00547.x. Epub 2010 May 18. PMID 20560997
- [Background] Gaskin EB, Levy S, Guzman-Armstrong S, Dawson D, Chalmers J. Knowledge, attitudes, and behaviors of federal service and civilian dentists concerning minimal intervention dentistry. Mil Med. 2010 Feb;175(2):115-21. doi: 10.7205/milmed-d-09-00140. PMID 20180481
- [Background] Shah AH, Sheddi FM, Alharqan MS, Khawja SG, Vohra F, Akram Z, Faden AA, Khalil HS. Knowledge and Attitude among General Dental Practitioners towards Minimally Invasive Dentistry in Riyadh and AlKharj. J Clin Diagn Res. 2016 Jul;10(7):ZC90-4. doi: 10.7860/JCDR/2016/20543.8207. Epub 2016 Jul 1. PMID 27630962
- [Background] Rayapudi J, Usha C. Knowledge, attitude and skills of dental practitioners of Puducherry on minimally invasive dentistry concepts: A questionnaire survey. J Conserv Dent. 2018 May-Jun;21(3):257-262. doi: 10.4103/JCD.JCD_309_17. PMID 29899626
- [Background] Riley JL 3rd, Qvist V, Fellows JL, Rindal DB, Richman JS, Gilbert GH, Gordan VV; DPBRN Collaborative Group. Dentists' use of caries risk assessment in children: findings from the Dental Practice-Based Research Network. Gen Dent. 2010 May-Jun;58(3):230-4. PMID 20478803
- [Background] Riley JL 3rd, Gordan VV, Ajmo CT, Bockman H, Jackson MB, Gilbert GH. Dentists' use of caries risk assessment and individualized caries prevention for their adult patients: Findings from The Dental Practice-Based Research Network. Tex Dent J. 2015 Jan;132(1):18-29. PMID 26234018
- [Background] Hurlbutt M, Young DA. A best practices approach to caries management. J Evid Based Dent Pract. 2014 Jun;14 Suppl:77-86. doi: 10.1016/j.jebdp.2014.03.006. Epub 2014 Mar 28. PMID 24929592
- [Background] [12] Afshar, M., khalafi, E., parizi, M., and Z. Shamsadini. 2019. Knowledge, Attitude and Practice Regarding Caries Risk Assessment and Management in General Dentists- A Cross Sectional SurveY, J. Evolution Med. Dent. Sci, Vol. 8, (3499-3504). (DOI;10. 14260/jemds/2019/757).